CLINICAL TRIAL: NCT01749644
Title: Switching From Tobramycin Inhalation Treatment to Tobramycin Inhaler Treatment: The Effect on CF Patients' Adherence and Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-12-9640-OE-CTIL
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Alteration in Quality of Life of CF Patients, Following Change of Treatment From Antibiotic Inhalation to Antibiotic Inhaler
Keywords: Cystic Fibrosis, Chronic Pseudomonas Infection, Inhaled Tobramycin
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CF patients with chronic pseudomonas infection

SUMMARY:
Pseudomonas is a common and virulent respiratory bacteria in patients with Cystic Fibrosis (CF). With time, the infection with Pseudomonas becomes chronic and very difficult to eradicate. The standard treatment of chronic Pseudomonas infection is inhaled Tobramycin which is given every other month.. Inhalation of Tobramycin was proven as an effective treatment that improves the respiratory function and reduces the concentration of bacteria in the sputum. However, inhaled treatment lasts between 15 to 30 minutes twice a day and therefore adherence is a major problem. The effect of switching from inhalation treatment to inhaler treatment on patient's adherence and quality of life has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years and above, Chronic Pseudomonas infection

Exclusion Criteria:

* Younger than 6 years; No chronic PSeudomonas infection

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CF patients with chronic pseudomonas infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in quality of life | 1 year

SECONDARY OUTCOMES:
Difference in exacerbation events | 1 year
  To be measured by:
  Worsening of CF symptoms such as coughing, sputum, deterioration in FEV1, all of which require hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ori Efrati, MD, Principal Investigator — Safra Children's hospital, National CF Center; Ifat Sarouk, MD, Principal Investigator — Safra Children's Hospital, National CF center
Locations (1):
- Safra Children's Hospital, Sheba Medical Center, Ramat Gan, Israel